CLINICAL TRIAL: NCT02760420
Title: Double-blind Randomized Controlled Clinical Trial of 3 Days of Amoxicillin Disperable Tablet (DT) Versus Placebo for Fast Breathing Childhood Pneumonia Among Children 2-59 Months of Age Presenting to Kamuzu Central Hospital in Lilongwe, Malawi
Brief Title: 3 Days Amoxicillin Versus Placebo for Fast Breathing Childhood Pneumonia in Malawi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Save the Children (Other)
Collaborators: University of North Carolina (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITIP1
Record Dates: First submitted 2016-05-01; First posted 2016-05-03 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): 250 mg of placebo (dispersible tablet) DT in two divided doses based on age bands (500 mg/day for children 2 months up to 12 months, 1000 mg/day for children 12 months up to 3 years, and 1,500 mg/day for children 3 years up to 5 years of age)
  Interventions: Drug: Placebo
- 3 Days (Active Comparator): 250 mg amoxicillin (dispersible tablet) DT in two divided doses based on age bands (500 mg/day for children 2 months up to 12 months, 1000 mg/day for children 12 months up to 3 years, and 1,500 mg/day for children 3 years up to 5 years of age)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Oral amoxicillin dispersible tablets (DT), 250 mg tablets, given according to age band, two times daily
  Arms: 3 Days
Drug: Placebo — Oral placebo dispersible tablets (DT), 250 mg tablets, given according to age band, two times daily
  Arms: Placebo

SUMMARY:
The purpose of this study to assess the effectiveness of no antibiotic treatment for fast breathing, community-acquired childhood pneumonia in a malaria-endemic region of Malawi.

ELIGIBILITY:
Inclusion Criteria:

* History of cough <14 days or difficult breathing with fast breathing (for children 2 to <12 months of age, >50 breaths/minute and for children >12 months of age, > 40 breaths/minute).
* Ability and willingness of children's caregiver to provide informed consent and to be available for follow-up for the planned duration of the study, including accepting a home visit if he/she fails to return to Kamuzu Central Hospital (KCH) with the child for a scheduled study follow-up visit.

Exclusion Criteria:

* If fast breathing observed at screening resolves after bronchodilator challenge.
* Chest-indrawing.
* Severe respiratory distress, classified by World Health Organization (WHO) pocketbook guidelines (e.g., grunting, nasal flaring, head nodding, crackles on auscultation, or very severe chest-indrawing).
* Presence of WHO Intergrated Management of Childhood Illness (IMCI) danger signs including: lethargy or unconsciousness, convulsions, vomiting everything, or inability to drink or breastfeed.
* Hypoxia (SaO2 < 90% on room air, as assessed by a Lifebox pulse oximeter).
* Stridor when calm.
* HIV-1 seropositivity or HIV-1 exposure, assessed as follows:

  * An HIV-positive result upon rapid antibody test will exclude any child from this study. If a child is less than 12 months or age or breastfeeding with a positive rapid test result, the child will be referred to receive additional confirmatory HIV testing (e.g., dried blood spot filter paper test) and follow-up from KCH staff, as per standard of care. Even if the confirmatory HIV testing subsequently shows that child is HIV-negative, he or she will remain excluded from the study.
  * If a child is less than 12 months of age or breastfeeding and has an HIV-negative result upon rapid antibody test, the child's biological mother's HIV status will need to be assessed. If the mother is HIV-positive, the child will be excluded. If the mother has a documented HIV-negative test result from within the past 3 months, the child will be included. If the mother does not have documentation of an HIV-negative test result, she will be tested via rapid antibody testing to determine the child's eligibility for this study.
  * If a child is over 12 months of age and not breastfeeding, an HIV-negative rapid antibody test is required for inclusion in the study.
  * Note: If a child has documentation of an HIV-negative test result from within the past 3 months, that test result will be used for the child's eligibility assessment.
* Severe acute malnutrition (weight for height/length < -3 SD, mid-upper arm circumference <115 mm, or edema).
* Possible tuberculosis (coughing for more than 14 days).
* Severe anemia, classified by WHO pocketbook guidelines (i.e., severe palmar pallor or hemoglobin <8.0 g/dL).
* Severe malaria, classified by WHO pocketbook guidelines (i.e., positive mRDT with any danger sign, stiff neck, abnormal bleeding, clinical jaundice, or hemoglobinuria).
* Known allergy to penicillin or amoxicillin.
* Receipt of an antibiotic treatment in the 48 hours prior to the study based on caregiver's self-report and/or documentation in child's medical record.
* Hospitalized within 14 days prior to the study.
* Living outside Lilongwe urban area, the study catchment area.
* Any medical or psychosocial condition or circumstance that, in the opinion of the investigators, would interfere with the conduct of the study or for which study participation might jeopardize the child's health.
* Any non-pneumonia acute medical illness which requires antibiotic treatment per local standard of care.
* Participation in a clinical study of another investigational product within 12 weeks prior to randomization or planning to begin participation during this study.
* Prior participation in an Innovative Treatments in Pneumonia study during a previous pneumonia diagnosis.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1126 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Proportion of children failing treatment | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ginsburg, MD, MPH, Principal Investigator — Consultant, University of Washington
Locations (2):
- Malawi (2):
  - Bwaila District Hospital, Lilongwe
  - Kamuzu Central Hospital, Lilongwe

REFERENCES:
- [Derived] Mvalo T, McCollum ED, Fitzgerald E, Kamthunzi P, Schmicker RH, May S, Phiri M, Chirombo C, Phiri A, Ginsburg AS. Chest radiography in children aged 2-59 months enrolled in the Innovative Treatments in Pneumonia (ITIP) project in Lilongwe Malawi: a secondary analysis. BMC Pediatr. 2022 Jan 10;22(1):31. doi: 10.1186/s12887-021-03091-3. PMID 35012490
- [Derived] May S, Brown SP, Schmicker RH, Emerson SS, Nkwopara E, Ginsburg AS. Non-inferiority designs comparing placebo to a proven therapy for childhood pneumonia in low-resource settings. Clin Trials. 2020 Apr;17(2):129-137. doi: 10.1177/1740774519888460. Epub 2019 Dec 8. PMID 31814441
- [Derived] Nkwopara E, Schmicker R, Mvalo T, Phiri M, Phiri A, Couasnon M, McCollum ED, Ginsburg AS. Analysis of serious adverse events in a paediatric fast breathing pneumonia clinical trial in Malawi. BMJ Open Respir Res. 2019 Sep 3;6(1):e000415. doi: 10.1136/bmjresp-2019-000415. eCollection 2019. PMID 31548894
- [Derived] Ginsburg AS, Mvalo T, Nkwopara E, McCollum ED, Ndamala CB, Schmicker R, Phiri A, Lufesi N, Izadnegahdar R, May S. Placebo vs Amoxicillin for Nonsevere Fast-Breathing Pneumonia in Malawian Children Aged 2 to 59 Months: A Double-blind, Randomized Clinical Noninferiority Trial. JAMA Pediatr. 2019 Jan 1;173(1):21-28. doi: 10.1001/jamapediatrics.2018.3407. PMID 30419120